CLINICAL TRIAL: NCT04329429
Title: An Open-label, Single-arm, Multi-center, Phase II Study of RC48-ADC in Subjects With HER2 Overexpressed Locally Advanced or Metastatic Biliary Tract Cancer (BTC) Who Have Failed First-line Chemotherapy
Brief Title: A Study of RC48-ADC in Subjects With HER2 Overexpressed Metastatic Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C010
Record Dates: First submitted 2020-03-27; First posted 2020-04-01 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC (Experimental): Participants will be treated with RC48-ADC 2.5 mg/kg, once every 2 weeks (Q2W) until investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or participant's decision to withdraw from therapy, or death (whichever occurs first)
  Interventions: Drug: RC48-ADC

INTERVENTIONS:
Drug: RC48-ADC — The eligible patients will be treated with RC48-ADC, an antibody-drug conjugate, 2.5 mg/kg, once every two weeks until investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or participant's decision to withdraw from therapy, or death (whichever occurs first)
  Other Names: Recombinant Humanized anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection

SUMMARY:
This study will evaluate the efficacy and safety of intravenous RC48-ADC in patients with locally advanced or metastatic HER2 overexpressed biliary tract cancer who have failed first-line chemotherapy.

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of intravenous RC48-ADC in patients with locally advanced or metastatic HER2 overexpressed biliary tract cancer who have failed first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years.
* Predicted survival ≥ 12 weeks.
* Diagnosed with histologically or cytologically-confirmed locally advanced or metastatic biliary tract cancer, including extra- or intra-hepatic bile duct cancer, gallbladder cancer, and ampulla cancer.
* Patients who have previously failed first-line chemotherapy. First-line chemotherapy failure is defined as disease progression (with imaging evidence of disease progression) during or within three months after treatment based on a two-drug combination of gemcitabine, platinum, or fluorouracil, or patients still cannot tolerate drug toxicity after two standardized drug reductions, or the disease progresses or relapses during neoadjuvant / adjuvant therapy or within six months after the end of treatment.
* At least one measurable lesion according to RECIST 1.1. The measurable lesion has not been treated with local treatment, including local radiotherapy, ablation and interventional treatment.
* HER2 overexpression (i.e. IHC 2+or 3+) as confirmed by the central laboratory. Subject is able to provide specimens from primary or metastatic lesions for HER2 tests.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function, evidenced by the following laboratory results:

Left ventricular ejection fraction ≥ 50 %. Hemoglobin (HGB) ≥ 90 g/L; WBC count≥ 3.0×10^9/L; Neutrophil count ≥ 1.5×10^9/L; Platelets ≥ 80×10^9/L.

Total bilirubin ≤ 1.5× ULN; AST and ALT ≤ 2.5×ULN or ≤ 5 x ULN with hepatic metastasis; Serum creatinine ≤1.5×ULN, or ≥ 50 ml/min of creatinine clearance (CrCl) according to Cockcroft-Gault formula.

* All female subjects will be considered to be of child-bearing potential unless they are postmenopausal, or have been sterilized surgically.Female subjects of child-bearing potential must agree to use at least one form of highly effective contraception. Female subjects must have serum pregnancy test negative within 7 days before study enrollment and must be non-lactating. Male subjects and their female partner who are of child-bearing potential must agree to use at least one form of highly effective contraception.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Received chemotherapy (treated with nitrosourea and mitomycin C within 6 weeks, oral fluorouracil within 2 weeks), radiotherapy (palliative local radiotherapy for bone metastases within 2 weeks before dosing), targeted therapy (the elution period of small molecule targeted drug is 2 weeks or 5 half-lives, whichever is longer), immunotherapy, or Chinese traditional medicine therapy (used Chinese traditional medicine with anti-tumor indications within one week) within 4 weeks before enrollment.
* Patients with biliary obstruction were excluded, unless the biliary obstruction was locally treated, such as endoscopic stent implantation, percutaneous liver puncture drainage, etc., with total bilirubin is reduced to 1.5 times of ULN.
* Have a history of malignancies other than biliary malignancies (except cured cervical carcinoma in situ or basal cell carcinoma of the skin and other malignancies that have been cured for 5 years).
* Previously received the treatment of other antibody-drug conjugates, e.g. T-DM1 and SGN-35.
* Have central nervous system (CNS) metastases and / or cancerous meningitis. Subjects who have received brain metastasis treatment may consider participating in this study, provided that the condition is stable for at least 6 months, and no disease progression has been confirmed by imaging examination within 4 weeks before administration, and all neurological symptoms have returned to baseline Level, no evidence of new or enlarged brain metastases, and discontinuation of radiation, surgery, or steroid treatment at least 28 days before the first dose of study treatment. This exception does not include cancerous meningitis, which should be ruled out regardless of its clinical status.
* Have severe, uncontrollable companion diseases, including combined uncontrollable infections, active tuberculosis, uncontrollable diabetes, and cardiovascular disease (New York Heart Association classification of Grade III or Grade IV heart failure, above Grade II cardiac conduction blockage, myocardial infarction, unstable arrhythmia or unstable angina in the past 12 months, cerebral infarction within 6 months, etc.), lung disease (History of interstitial pneumonia, obstructive pulmonary disease, and symptomatic bronchi spasm), deep vein thrombosis or pulmonary embolism within 12 months, decompensated liver cirrhosis.
* Have active autoimmune diseases that require systemic treatment (such as disease-modifying drugs, corticosteroids, or immunosuppressive drugs) in the past 2 years, the related alternative treatments (such as thyroxine, insulin, or adrenal or pituitary insufficiency corticosteroid replacement therapy) are permitted.
* Toxicity of previous anti-tumor treatment not recovered to CTCAE Grade 0-1 (with exception of Grade 2 alopecia), except for those who have hair loss, pigmentation, anemia, weakness and those who cannot recover from the long-term toxicity caused by radiotherapy.
* HIV positive; HBsAg positive with HBV-DNA positive (≥2000 copies/ml); HCV positive, except for patients with HCV positive and HCV-RNA negative in PCR test.
* History of major surgery within 4 weeks of planned start of trial treatment, or patients with previous allogeneic hematopoietic stem cell transplant or organ transplant.
* Has received anti-cancer vaccine within 4 weeks of planned start of trial treatment, or planned to receive anti-cancer vaccine during trial treatment.
* Pleural or abdominal effusion with clinical symptoms that requires ongoing treatment.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Duration of Objective Response (DOR) | 24 months
  DOR was defined as the time from first documented OR to first documented PD or death from any cause, whichever occurred earlier
Progression Free Survival (PFS) | 24 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Overall Survival(OS) | Up to 24 months
  OS was defined as the time from the first study treatment to the date of death from any cause.
Disease control rate (DCR) | 24 months
  DCR was defined as the proportion of patients who achieved an objective response or maintained stable disease
Adverse Events | 28 days after the last dose of study treatment
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Fang, Ph.D, Study Director — RemeGen Co., Ltd.
Locations (16):
- China (16):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beijing 302 Hospital/5th Medical Center of Chinese PLA General of Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality
  - The First Hospital Affiliated to AMU (Southwest Hospital), Chongqing, Chongqing Municipality
  - Sun Yat-Sen university Cancer Center, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan
  - First Hospital of Jilin University, Changchun, Jilin
  - Shandong Cancer Hospital Affiliated to Shandong University, Jinan, Shandong
  - Eastern Hepatobiliary Surgery Hospital, Second Military Medical University, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tongji University Shanghai East Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No